CLINICAL TRIAL: NCT05787379
Title: Leveraging Knowledge of Chronic Multisymptom Illness to Improve Care for Veterans
Brief Title: Care for Veterans Post-COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDR 23-001
Record Dates: First submitted 2023-03-23; First posted 2023-03-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: training; COVID-19; post-acute sequelae of COVID infection
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: The Concordant Care approach involves engaging in processes that: 1) validate the patient's experience, 2) develop a shared understanding of the condition, and 3) create a patient-centered, whole health-oriented action plan to manage the condition. The training involves four components: completion of approx. 3 hours of online, asynchronous training; attendance to at least two tele-mentoring sessions to review specific cases, didactics, role-play exercises, and session recordings; obtaining a clinician pocket care with reminders of Concordant Care process; and being prompted by a Veteran patient to talk about their concerns with Long-COVID.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Providers receiving Long-COVID Concordant Care Training (Experimental): Providers randomized to this arm will receive concordant care training.
  Interventions: Behavioral: Concordant Care Training
- Providers receiving Education Packet Training (Active Comparator): Providers randomized to this arm will receive education packet training.
  Interventions: Behavioral: Education Packet Training

INTERVENTIONS:
Behavioral: Concordant Care Training — Concordant Care training has four components. 1. Clinicians will complete ~3 hours of online, asynchronous training that will teach them practices including validate Veterans' experiences with Long-COVID, develop shared understanding with patients about Long-COVID, and develop patient-centered action plans. Clinicians will be provided with handouts, case examples, video demonstrations, and practice exercises to help them integrate these practices into care. 2. Tele-mentoring groups will be offered ~bi-weekly and be open to all clinician participant in the Concordant Training arm. Content will include review of specific cases, didactics on specific Concordant Care practices, role-play exercises, and review of session recordings. At least two sessions are required. 3. Clinician Pocket Card that serves as a reminder of the Concordant Care process. 4. An electronic prompt will be sent to enrolled Veterans encouraging them to speak with their clinician about their Long-COVID concerns.
  Arms: Providers receiving Long-COVID Concordant Care Training
Behavioral: Education Packet Training — Clinicians randomized to the control arm will receive a comprehensive information packet with the latest understanding of Long-COVID. Clinicians will also be provided a packet directing them to relevant VA trainings for Long-COVID. Whole Health trainings which focus on wholistic integrated approaches to care will be highlighted. Whole Health is important for all Veterans, and it is thought to be particularly relevant for poorly understood conditions that don't easily fit in traditional medical model.
  Arms: Providers receiving Education Packet Training

SUMMARY:
The evidence-based Concordant Care approach involves engaging in processes that: 1) validate the patient's experience, 2) develop a shared understanding of the condition, and 3) create a patient-centered, whole health-oriented action plan to manage the condition. This is consistent with published expert opinion that Concordant Care underlies patients' (and clinicians') positive experiences of care for poorly understood conditions. Despite strong evidence supporting this care approach, there are no interventions to train clinicians on practices to provide Concordant Care for Veterans with poorly understood conditions such as Long-COVID. Part 1 of the study will optimize and test if a Concordant Care training improves VA clinicians' engagement in recommended practices to provide Concordant Care (i.e., validate, shared understanding, action plan) for Veterans with Long-COVID. This study will adapt and refine Concordant Care training for Long-COVID. Part 2 of this study will determine if Concordant Care training increases clinicians' engagement in recommended practices to provide Concordant Care and will explore the effectiveness of Concordant Care on care outcomes including satisfaction, adherence to care, & disability for Veterans with Long-COVID. Veterans treated by clinicians receiving Concordant Care training will report their clinician more frequently engaged in recommended conversations (i.e., ask about Long-COVID, validate experience with Long-COVID, create a shared understanding and action plan), and Veterans will perceive greater shared understanding of Long-COVID with their clinicians than Veterans treated by clinicians in the control arm.

DETAILED DESCRIPTION:
This is a two-part study. Part 1 of the study will optimize and test if a Concordant Care training improves VA clinicians' engagement in recommended practices to provide Concordant Care (i.e., validate, shared understanding, action plan) for Veterans with Long-COVID. The evidence-based Concordant Care approach involves engaging in processes that: 1) validate the patient's experience, 2) develop a shared understanding of the condition, and 3) create a patient-centered, whole health-oriented action plan to manage the condition. Concordant Care will be adapted through interviews and focus groups with Veterans with Long-COVID (estimated n=9) and primary care providers (estimated n=21). Feedback from the participants will help refine and test Concordant Care training. Part 2 of this study will determine if Concordant Care training increases clinicians' engagement in recommended practices to provide Concordant Care and will explore the effectiveness of Concordant Care on care outcomes including satisfaction, adherence to care, & disability for Veterans with Long-COVID. Part 2 will be a randomized parallel cluster trial with primary care clinicians (n=60) separated into a Concordant Care training group and an education packet control group. Veterans (n=240) who have an upcoming appointment with their primary care provider who is a participant in the study will be recruited. The Veterans will be assessed at baseline before their appointment and approximately 3-months later after their appointment. Veterans treated by clinicians receiving Concordant Care training will report their clinician more frequently engaged in recommended conversations (i.e., ask about Long-COVID, validate experience with Long-COVID, create a shared understanding and action plan), and Veterans will perceive greater shared understanding of Long-COVID with their clinicians than Veterans treated by clinicians in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 and Part 2, English-speaking VA primary care providers will be included.
* Part 1, Veterans who self-identify as having Long-COVID will be included.
* Part 2, Veterans who meet criteria for Long-COVID assessed with modified DePaul Symptom Questionnaire version 2 will be included;
* Part 2, Veterans must also have a scheduled appointment with one of the participating clinicians within one to six months of the clinician being consented.

Exclusion Criteria:

* Part 1 and Part 2, clinicians who have already taken Concordant Care training will be excluded.
* Part 1, Veterans will be excluded if they are not receiving care in the VA.
* Part 2, Veterans will be excluded if they were in the Intensive Care Unit (ICU) for COVID-19.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Concordant Care Practice Change | Baseline and 3-months
  Concordant Care practices will be measured with the 11-item measure that asks the patient if the clinician talked with them about multiple dimensions of their understanding of the health condition (i.e., cause, consequence, treatment). Participants answer yes or no to each question. Scores range from 0 to 11 with a higher score = more Concordant Care practices.
Concordance of Illness Perceptions Questionnaire Change | Baseline and 3-months
  Shared Understanding will be captured with the concordance of illness perceptions questionnaire, a 6-item validated measure of shared understanding of the 5 components of illness perception between patients and clinicians. Veterans respond on a 5-point Likert scale. Scores range from 6 to 30 with higher scores = greater concordant understanding.

SECONDARY OUTCOMES:
Patient Satisfaction Questionnaire (PSQ-III) | Baseline and 3-months
  The 18-item PSQ measures patient satisfaction in health care services and has been used specifically to assess patient satisfaction of VA healthcare services. Response options are 1-5 with 1=strongly agree and 5=strongly disagree. Scores range from 18 to 90 with higher scores = greater satisfaction with medical care.
Medical Outcomes Survey Adherence Scale | Baseline and 3-months
  The Medical Outcomes Survey Adherence 5-item scale captures Veterans adherence to primary care clinician's recommendations. Scores range from 6 to 30 with greater scores = better adherence.
Veterans Rand (VR-12) | Baseline and 3-months
  Veterans Rand 12-item Health Survey (VR-12). The VR-12 is a well-validated quality of life measure that assesses multiple domains of physical and mental health functioning. Scores range from 0 to 100 with higher scores = less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marie McAndrew, PhD, Principal Investigator — East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ
Locations (1):
- East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No